CLINICAL TRIAL: NCT01601821
Title: An Open Label Comparative Study Of De Novo Renal Allograft Recipients Receiving CSA + MMF + Corticosteroids Versus CSA + Rapamune + Corticosteroids With Further CSA Elimination In The Rapamune Arm With The Introduction Of MMF
Brief Title: Open Label Comparative Study Of De Novo Renal Allograft Recipients Receiving CSA + MMF + Corticosteroids Versus CSA + Rapamune + Corticosteroids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468H-102012; B1741220
Record Dates: First submitted 2012-05-03; First posted 2012-05-18 (Estimated); Results first posted 2013-06-19 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-11

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (CsA+Rapamune+CS) (Active Comparator)
  Interventions: Drug: CsA+Rapamune+CS
- Arm B (CsA+MMF+CS) (Experimental)
  Interventions: Drug: CsA+MMF+CS

INTERVENTIONS:
Drug: CsA+Rapamune+CS — Part 1: Rapamune will be given as a loading dose of 6 mg once followed by maintenance dose of 2 mg to achieve a target trough level of 8-15 ng/ml. Part 2: Rapamune dose will be adjusted to achieve a target trough level of 10-15ng/ml through 6 months
  Arms: Arm A (CsA+Rapamune+CS)
Drug: CsA+MMF+CS — The control arm is the standard local practice (official protocol) in Iran:
  Cyclosporine + MMF + Corticosteroid. The time period is from pre-study screening / baseline evaluation up to 12 months for patients who are maintained on CsA + MMF + CS.
  Arms: Arm B (CsA+MMF+CS)

SUMMARY:
To compare the safety and efficacy of cyclosporine (CsA) + mycophenolate mofetil (MMF) + corticosteroids © to CsA + Rapamune + Cs with CsA elimination in the Rapamune arm with the introduction of MMF in de novo renal allograft recipients.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 years and weight 40 kg
* End-stage renal disease, with patients receiving a primary or secondary renal allograft from a living-unrelated donor, or from a living-related donor.
* Women who are of childbearing potential must have a negative pregnancy test before enrollment in the study and agree to use a medically acceptable method of contraception throughout the treatment period and for 3 months following discontinuation from the study.
* Total white blood cell count 4.0 x 109/L (4,000/mmP3P), platelet count 100 x 10P9P/L(100,000/mmP3P), fasting triglycerides ≤ 4.6 mmol/L (400 mg/dL), fasting cholesterol ≤ 7.8 mmol/L (300 mg/dL). If it is not possible to obtain fasting triglycerides and cholesterol before surgery, historical values (within 1 year) may be used.
* Signed and dated informed consent (parent or legal guardian must provide consent for patients <18 years of age). An assent form will be signed by patients < 18 years of age enrolled in the study.

Exclusion Criteria:

* Evidence of active systemic or localized major infection at the time of initial Sirolimus administration.
* Cadaveric donors
* History of malignancy within 5 years before enrollment into the study (with the exception of adequately treated basal cell or squamous cell carcinoma of the skin)
* Use of any investigational drug other than specified in the protocol during the 4 weeks before enrolling in the study.
* Use of planned antibody induction therapy at the time of transplantation.
* Active gastrointestinal disorder that may interfere with drug absorption.
* Known hypersensitivity to Sirolimus, MMF or Cyclosporine or its derivatives.
* Multiple organ transplants (2 or more organ transplant e.g. Kidney and Pancreas).
* Patient with high risk of rejection (eg. Patients with a PRA >50%, black patients and patients with 2nd transplant who lost their first graft within the first 6 months).
* Evidence of infiltrate, cavitation, or consolidation on chest x-ray obtained during pre-study screening

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 245 (Actual)
Dates: Start 2006-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Iran (4):
  - Labbafinejad Hospital, Tehran
  - Modarres Hospital, Tehran
  - Shariati Hospital, Tehran
  - Taleqani Hospital, Tehran

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0468H-102012

RESULTS

PARTICIPANT FLOW:
Groups:
- CsA+Rapamune+CS: Month 0-3: rapamune 6 milligram (mg) tablet orally once as a loading dose within 48 hours of transplantation, followed by rapamune 2 mg tablet orally once daily as a maintenance dose to achieve a target trough level of 8-15 nanogram per milliliter (ng/mL) in combination with cyclosporine (CsA) tablets orally to achieve a trough level of 150-250 ng/mL. Month 4-6: CsA was withdrawn abruptly, mycophenolate mofetil (MMF) tablet orally at a dose of 1-1.5 grams per day (g/day) and rapamune dose adjusted to achieve a target trough level of 10-15 ng/mL. Month 7-12: rapamune dose adjusted to achieve a target trough level of 8-12 ng/mL, MMF tablet orally at a dose of 1-1.5 g/day. Participants also received corticosteroids (CS) tablets orally as per local practice with a minimum daily dose of 5 mg over 12 months.
- CsA+MMF+CS: Month 0-5: CsA tablets orally to achieve a trough level of 150-300 ng/mL. Month 6-12: CsA tablets orally to achieve a trough level of 100-200 ng/mL. Participants also received MMF tablet orally at a dose of 2 g/day and CS tablets orally as per local practice with a minimum daily dose of 5 mg over 12 months.
Period: Overall Study
Arm/Group | CsA+Rapamune+CS | CsA+MMF+CS
Started | 125 | 120
Completed | 96 | 91
Not Completed | 29 | 29
Not completed — Death | 2 | 5
Not completed — Protocol Violation | 2 | 2
Not completed — Lost to Follow-up | 6 | 14
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Graft Loss | 6 | 6
Not completed — Study Events | 7 | 1
Not completed — Other | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- CsA+Rapamune+CS: Month 0-3: rapamune 6 mg tablet orally once as a loading dose within 48 hours of transplantation, followed by rapamune 2 mg tablet orally once daily as a maintenance dose to achieve a target trough level of 8-15 ng/mL in combination with CsA tablets orally to achieve a trough level of 150-250 ng/mL. Month 4-6: CsA was withdrawn abruptly, MMF tablet orally at a dose of 1-1.5 g/day and rapamune dose adjusted to achieve a target trough level of 10-15 ng/mL. Month 7-12: rapamune dose adjusted to achieve a target trough level of 8-12 ng/mL, MMF tablet orally at a dose of 1-1.5 g/day. Participants also received CS tablets orally as per local practice with a minimum daily dose of 5 mg over 12 months.
- Total: Total of all reporting groups
Arm/Group | CsA+Rapamune+CS | CsA+MMF+CS | Total
Number analyzed (Participants) | 125 | 120 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (13.4) | 41.6 (15.1) | 39.9 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 45 | 92
  Male | 78 | 75 | 153

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Efficacy Failure
Description: Efficacy failure was defined as first occurrence of either biopsy confirmed acute rejection, graft loss or death within 12 months of post-transplantation. Percentage of participants with efficacy failure was reported.
Time Frame: Baseline up to Month 12
Population: Per-protocol 1 (PP1) population included all participants who had completed study, also included those who dropped out of study due to occurrence of death, graft loss, or biopsy-confirmed acute rejection and had no major protocol deviations.
Measure: Number; unit: percentage of participants
Arm/Group | CsA+Rapamune+CS | CsA+MMF+CS
Number analyzed (Participants) | 105 | 104
percentage of participants | 11.4 | 13.5
Statistical Analysis 1: Comparison: CsA+Rapamune+CS vs CsA+MMF+CS; Chi-square test was used to test superiority of arm CsA+Rapamune+CS versus arm CsA+MMF+CS; Test type: Superiority or Other; p = 0.341, Chi-squared; percent difference = -2.0, 90% CI 2-sided [-5.5 to 1.5]

2. Secondary Outcome: Serum Creatinine Level
Description: Serum creatinine is an indicator of kidney function. Creatinine is a substance formed from the metabolism of creatine, commonly found in blood, urine and muscle tissue. It is removed from the blood by the kidneys and excreted in urine. An increased level of creatinine in the blood indicates decreased kidney function. Normal adult blood levels of creatinine are 0.5 to 1.1 milligram per deciliter (mg/dL) for females and 0.6 to 1.2 mg/dL for males; however, the normal values are age-dependent as elderly patients typically have smaller muscle mass.
Time Frame: Month 3, 6, 12
Population: PP1 population. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' is number of participants evaluable at specific time points for each arm group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CsA+Rapamune+CS | CsA+MMF+CS
Number analyzed (Participants) | 102 | 94
mg/dL
  Month 3 (n=102, 94) | 1.4 (0.4) | 1.4 (0.4)
  Month 6 (n=101, 92) | 1.2 (0.3) | 1.3 (0.4)
  Month 12 (n=98, 91) | 1.2 (0.3) | 1.3 (0.3)
Statistical Analysis 1: Comparison: CsA+Rapamune+CS vs CsA+MMF+CS; Month 3: One-way analysis of variance (ANOVA) was used to test the difference; Test type: Superiority or Other; p = 0.870, ANOVA — Statistical testing was based on 5% significance level
Statistical Analysis 2: Comparison: CsA+Rapamune+CS vs CsA+MMF+CS; Month 6: One-way ANOVA was used to test the difference; Test type: Superiority or Other; p = 0.381, ANOVA — Statistical testing was based on 5% significance level
Statistical Analysis 3: Comparison: CsA+Rapamune+CS vs CsA+MMF+CS; Month 12: One-way ANOVA was used to test the difference; Test type: Superiority or Other; p = 0.096, ANOVA — Statistical testing was based on 5% significance level

3. Secondary Outcome: Creatinine Clearance
Description: Creatinine clearance (CCr) is a measure of kidney function. CCr is the volume of blood plasma that is cleared of creatinine by the kidneys per unit time. Normal values for healthy, young males are in the range of 100-135 millimeters per minute (mL/min) and for females, 90-125 mL/min. Creatinine clearance decreases with age. A low creatinine clearance rate indicates poor kidney function.
Time Frame: Month 3, 6, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | CsA+Rapamune+CS | CsA+MMF+CS
Number analyzed (Participants) | 102 | 94
mL/min
  Month 3 (n=102, 94) | 64.0 (19.9) | 63.9 (16.0)
  Month 6 (n=101, 92) | 72.8 (19.3) | 71.6 (18.3)
  Month 12 (n=98, 91) | 76.4 (22.7) | 74.0 (28.6)
Statistical Analysis 1: Comparison: CsA+Rapamune+CS vs CsA+MMF+CS; Month 3: One-way ANOVA was used to test the difference; Test type: Superiority or Other; p = 0.979, ANOVA — Statistical testing was based on 5% significance level
Statistical Analysis 2: Comparison: CsA+Rapamune+CS vs CsA+MMF+CS; Month 6: One-way ANOVA was used to test the difference; Test type: Superiority or Other; p = 0.660, ANOVA — Statistical testing was based on 5% significance level
Statistical Analysis 3: Comparison: CsA+Rapamune+CS vs CsA+MMF+CS; Month 12: One-way ANOVA was used to test the difference; Test type: Superiority or Other; p = 0.518, ANOVA — Statistical testing was based on 5% significance level

4. Secondary Outcome: Glomerular Filtration Rate (GFR) by Nankivell Method
Description: GFR is an index of kidney function. GFR describes the flow rate of filtered fluid through the kidney. GFR was calculated using the Nankivell formula. GFR by Nankivell equation= (6.7 per serum creatinine) plus (0.25*body weight) minus (0.5*serum urea) minus (100 per height square) plus (35 for male or 25 for female). A normal GFR is greater than (>)90 mL/min per 1.73 m^2 [mL/min/1.73 m^2], although children and older people usually have a lower GFR. Lower values indicated poor kidney function. A GFR less than (<)15 mL/min/1.73 m^2 indicated kidney failure.
Time Frame: Month 3, 6, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | CsA+Rapamune+CS | CsA+MMF+CS
Number analyzed (Participants) | 102 | 94
mL/min/1.73 m^2
  Month 3 (n=102, 94) | 59.5 (20.4) | 58.8 (15.2)
  Month 6 (n=101, 92) | 65.2 (16.0) | 64.3 (19.5)
  Month 12 (n=98, 91) | 67.4 (17.5) | 67.5 (46.5)
Statistical Analysis 1: Comparison: CsA+Rapamune+CS vs CsA+MMF+CS; Month 3: One-way ANOVA was used to test the difference; Test type: Superiority or Other; p = 0.786, ANOVA — Statistical testing was based on 5% significance level
Statistical Analysis 2: Comparison: CsA+Rapamune+CS vs CsA+MMF+CS; Month 6: One-way ANOVA was used to test the difference; Test type: Superiority or Other; p = 0.738, ANOVA — Statistical testing was based on 5% significance level
Statistical Analysis 3: Comparison: CsA+Rapamune+CS vs CsA+MMF+CS; Month 12: One-way ANOVA was used to test the difference; Test type: Superiority or Other; p = 0.977, ANOVA — Statistical testing was based on 5% significance level

5. Secondary Outcome: Incidence of Biopsy-Confirmed Acute Rejection
Description: Diagnosis of acute rejection was made via kidney biopsy using Banff criteria. Percentage of participants with biopsy-confirmed acute rejection was reported.
Time Frame: Baseline up to Month 6
Population: PP2 population included all participants who had completed study, also included those who dropped out of the study due to biopsy confirmed acute rejection at Month 6.
Measure: Number; unit: percentage of participants
Arm/Group | CsA+Rapamune+CS | CsA+MMF+CS
Number analyzed (Participants) | 100 | 95
percentage of participants | 4.0 | 3.2
Statistical Analysis 1: Comparison: CsA+Rapamune+CS vs CsA+MMF+CS; Fisher's exact test was used to test the difference; Test type: Superiority or Other; p = 0.999, Fisher Exact — Statistical testing was based on 5% significance level

6. Secondary Outcome: Histologic Grade of First Acute Rejection
Description: Diagnosis of acute rejection was made via kidney biopsy. Categorization of biopsies with suspected acute rejection was based on histological findings using updated 1997 Banff criteria. Grade 1A: cases with significant interstitial infiltration (>25% of parenchyma affected) and foci of moderate tubulitis (5-10 cells/tubular cross section), Grade 1B: with severe tubulitis (>10 cells/tubular cross section), Grade 2A: mild-moderate intimal arteritis, Grade 2B: severe intimal arteritis and Grade 3: transmural arterits and/or fibrinoid necrosis. Data is reported as percentage of participants.
Time Frame: Baseline up to Month 12
Population: PP2 population included all participants who had completed study, also included those who dropped out of the study due to biopsy confirmed acute rejection at Month 6. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | CsA+Rapamune+CS | CsA+MMF+CS
Number analyzed (Participants) | 3 | 3
percentage of participants
  1A | 100.0 | 66.7
  1B | 0.0 | 33.3

7. Secondary Outcome: Percentage of Participants Who Survived
Description: Survival defined as participants living with or without a functioning graft.
Time Frame: Month 12
Population: PP3 population included all participants who had completed study, also included those who dropped out of the study due to the occurrence of death.
Measure: Number; unit: percentage of participants
Arm/Group | CsA+Rapamune+CS | CsA+MMF+CS
Number analyzed (Participants) | 98 | 96
percentage of participants | 98.0 | 94.8
Statistical Analysis 1: Comparison: CsA+Rapamune+CS vs CsA+MMF+CS; Fisher's exact test was used to test the difference; Test type: Superiority or Other; p = 0.276, Fisher Exact — Statistical testing was based on 5% significance level

8. Secondary Outcome: Percentage of Participants With Graft Survival
Description: Graft survival defined as those participants who did not experience graft loss. Graft loss defined as physical loss (nephrectomy), functional loss (necessitating maintenance dialysis for >8 weeks), retransplant or death during the first 12 months after randomization.
Time Frame: Month 12
Population: PP4 population included all participants who had completed study, also included those who dropped out of the study due to the occurrence of graft loss.
Measure: Number; unit: percentage of participants
Arm/Group | CsA+Rapamune+CS | CsA+MMF+CS
Number analyzed (Participants) | 102 | 97
percentage of participants | 94.1 | 93.8
Statistical Analysis 1: Comparison: CsA+Rapamune+CS vs CsA+MMF+CS; Fisher's exact test was used to test the difference; Test type: Superiority or Other; p = 0.999, Fisher Exact — Statistical testing was based on 5% significance level

9. Secondary Outcome: Incidence of Presumptive or Documented Infection
Description: Presumptive or documented infection during the 12 months after transplantation; was confirmed by culture, biopsy, or serology and reported. Percentage of participants with presumptive or documented infection was reported.
Time Frame: Baseline up to Month 12
Population: Analysis population included all participants enrolled in the study. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | CsA+Rapamune+CS | CsA+MMF+CS
Number analyzed (Participants) | 123 | 118
percentage of participants | 20.3 | 18.6
Statistical Analysis 1: Comparison: CsA+Rapamune+CS vs CsA+MMF+CS; Chi-square test was used to test the difference; Test type: Superiority or Other; p = 0.868, Chi-squared — Statistical testing was based on 5% significance level

10. Secondary Outcome: Incidence of Histologically Confirmed Lymphoproliferative Disease
Description: Lymphoproliferative disorder represents an abnormal proliferation of B cells in response to either primary or reactivated infection with Epstein-Barr virus. Percentage of participants with histologically confirmed lymphoproliferative disease was reported.
Time Frame: Baseline up to Month 12
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | CsA+Rapamune+CS | CsA+MMF+CS
Number analyzed (Participants) | 97 | 91
percentage of participants | 1.0 | 0.0
Statistical Analysis 1: Comparison: CsA+Rapamune+CS vs CsA+MMF+CS; Fisher's exact test was used to test the difference; Test type: Superiority or Other; p = 0.999, Fisher Exact — Statistical testing was based on 5% significance level

11. Secondary Outcome: Percentage of Participants With Efficacy Failure or Premature Elimination
Description: Efficacy failure was defined as the first occurrence of acute rejection, graft loss, or death. Premature elimination was defined as elimination from the study for any other reason.
Time Frame: Month 12
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | CsA+Rapamune+CS | CsA+MMF+CS
Number analyzed (Participants) | 123 | 118
percentage of participants | 22.0 | 22.9
Statistical Analysis 1: Comparison: CsA+Rapamune+CS vs CsA+MMF+CS; Chi-square test was used to test the difference; Test type: Superiority or Other; p = 0.985, Chi-squared — Statistical testing was based on 5% significance level

12. Secondary Outcome: Incidence of Anemia
Description: Diagnostic criterion for anemia was based on the laboratory results; in men: hemoglobin (Hb) <14 gram per deciliter (g/dL), hematocrit (Hct) <42%, or red blood cells (RBCs) <4.5 million/liter (million/L); for women: Hb <12 g/dL, Hct <37%, or RBC < 4 million/L. Percentage of participants with anaemia was reported.
Time Frame: Baseline up to Month 12
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | CsA+Rapamune+CS | CsA+MMF+CS
Number analyzed (Participants) | 123 | 118
percentage of participants | 94.3 | 98.3
Statistical Analysis 1: Comparison: CsA+Rapamune+CS vs CsA+MMF+CS; Fisher's exact test was used to test the difference; Test type: Superiority or Other; p = 0.172, Fisher Exact — Statistical testing was based on 5% significance level

13. Secondary Outcome: Number of Participants Who Discontinued
Description: Number of participants who discontinued the study treatment due to any reason is reported.
Time Frame: Month 12
Population: Analysis population included all participants enrolled in the study.
Measure: Number; unit: participants
Arm/Group | CsA+Rapamune+CS | CsA+MMF+CS
Number analyzed (Participants) | 125 | 120
participants | 29 | 29
Statistical Analysis 1: Comparison: CsA+Rapamune+CS vs CsA+MMF+CS; Chi-square test was used to test the difference; Test type: Superiority or Other; p = 0.978, Chi-squared — Statistical testing was based on 5% significance level

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CsA+Rapamune+CS | CsA+MMF+CS
Serious Adverse Events (participants affected / at risk) | 56/125 | 44/120
Other Adverse Events (participants affected / at risk) | 67/125 | 44/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CsA+Rapamune+CS (N=125) | CsA+MMF+CS (N=120)
Aplasia pure red cell (Blood and lymphatic system disorders) | 2 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 4 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 0
Gastroenteritis (Gastrointestinal disorders) | 4 | 1
Volvolus (Gastrointestinal disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Peripheral oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Transplant rejection (Immune system disorders) | 13 | 10
Candidiasis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 5
Diabetic foot infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 1
Lung infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1
Penile infection (Infections and infestations) | 0 | 1
Perlvic abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 1 | 3
Sepsis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 8 | 3
Wound infection (Infections and infestations) | 4 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 2 | 0
Kidney rupture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Postoperative wound complications (Injury, poisoning and procedural complications) | 0 | 2
Seroma (Injury, poisoning and procedural complications) | 1 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 6 | 4
Blood creatinine increased (Investigations) | 17 | 5
Blood glucose increased (Investigations) | 1 | 1
Blood urea increased (Investigations) | 1 | 0
Cytomegalovirus test positiv (Investigations) | 1 | 4
Lipids increased (Investigations) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 3
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Hyperoxaluria (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Renal artery thrombosis (Renal and urinary disorders) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 3 | 3
Ureteral necrosis (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 2
Ureteric stenosis (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arterial thrombosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Lymphocele (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CsA+Rapamune+CS (N=125) | CsA+MMF+CS (N=120)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 5 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 0
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Oral disorder (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Peripheral oedema (General disorders) | 2 | 0
Transplant rejection (Immune system disorders) | 2 | 1
Candidiasis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 3
Fungal infection (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Oral infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 5
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 2 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 3 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 7 | 4
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood cholesterol increased (Investigations) | 11 | 3
Blood creatinine increased (Investigations) | 4 | 6
Blood glucose increased (Investigations) | 6 | 5
Blood triglycerides increased (Investigations) | 15 | 5
Cytomegalovirus test positive (Investigations) | 2 | 4
Drug level increased (Investigations) | 2 | 0
Haemoglobin decreased (Investigations) | 6 | 6
Immunosuppressant drug level increased (Investigations) | 0 | 1
Lipids increased (Investigations) | 2 | 0
Liver function test abnormal (Investigations) | 21 | 8
Platelet count decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Delirium (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 3 | 2
Renal vein thrombosis (Renal and urinary disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Lymphocele (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.